CLINICAL TRIAL: NCT03708094
Title: A Study for Predicting the Prognosis of Renal Transplantation by the Clear Pathogenic Gene of End-stage Renal Disease in Children
Brief Title: Prognosis Study of Renal Transplantation in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Boston Children's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Central South University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Hong Xu，MD.PhD, Professor, Children's Hospital of Fudan University
Other Study IDs: TxGene 1.0
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Kidney Failure
Keywords: prognosis; pathogenic gene; decision tree study
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- molecular diagnosis confirmed: Whole exome sequencing is applied to children and the molecular diagnosis was identified before renal transplantation.
  Interventions: Diagnostic Test: molecular diagnosis
- molecular diagnosis unconfirmed: Whole exome sequencing is applied to children and the molecular diagnosis was not identified before renal transplantation.

INTERVENTIONS:
Diagnostic Test: molecular diagnosis — whole exome sequencing and data analysis to elucidating molecular diagnosis
  Groups: molecular diagnosis confirmed

SUMMARY:
Kidney transplantation is the worldwide recognized best renal replacement treatment for children with end-stage renal disease. Successful kidney transplantation can not only alleviate uremia symptoms, improve survival and quality of life, but also achieve optimal growth and cognitive development in children. Clarifying the cause of end-stage renal disease before transplantation is of vital importance to the comprehensive assessment and follow-up of the extra renal organs, reducing the risk of recurrence of the primary disease, the choice of the timing and the mode of transplantation, the scheme of immunosuppressive agents, as well as providing accurate genetic counseling for families. Timely molecular diagnosis and correct data analysis play a positive role in promoting the etiological diagnosis of uremic children before renal transplantation. We hypothesized that identifying the molecular diagnosis can improve prognosis of kidney transplantation. 300 cases of end-stage renal disease children were included and whole exome sequencing are performed to identify the molecular diagnosis. The cohort was divided into 2 groups according to whether the molecular diagnosis was clear. Clinical information before and after renal transplantation of each group are collected, and the decision tree analysis model and logistic regression model are used to study the effect of clear molecular diagnosis on the 3 year survival rate of renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Donors and recipients who accepted kidney transplantation at centers included in this study

Exclusion Criteria:

* Older than 18 years old.
* There are severe systemic diseases and/or local and/or spiritual system diseases.
* There are systemic acute or chronic infections, infectious diseases.
* The donated organ dysfunction, or other causes that are damage to donors and recipients.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 300 continuous renal transplant cases from multiple centers included in this study
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Renal graft survival rate | 3 years after renal transplantation
  The number of survival renal transplant graft in the 3 year observation period accounted for the percentage of the total cases studied.

SECONDARY OUTCOMES:
Incidence of acute rejection | 3 years after renal transplantation
  The number of acute rejection after transplantation during the 3 year observation period accounted for the percentage of the total cases studied.
Recurrence rate of primary disease | 3 years after renal transplantation
  The number of patient with primary disease recurrence during the 3 year observation period accounted for the percentage of the total cases studied.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, MD.PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No